CLINICAL TRIAL: NCT06575556
Title: Validation of Magnetic Resonance Imaging Against Multidetector Computed Tomography After Ross Procedure Using Loose Jacket Technique
Brief Title: Validation of MRI Instead of CT to Follow-up Ross Procedure With Loose Jacket Technique
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Gamal Ahmed Ramadan, Doctor, Assiut University
Other Study IDs: MRI in Ross procedure
Record Dates: First submitted 2024-07-13; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Imaging
Keywords: Cardiac imaging; Cardiac CT; Cardiac MRI; Ross procedure; Loose jacket technique
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent Ross procedure with loose jacket technique: Patients who underwent Ross procedure with loose jacket technique regardless of the timing of surgery, all patients will undergo both CT and MRI scans
  Interventions: Diagnostic Test: Cardiac CT and MRI

INTERVENTIONS:
Diagnostic Test: Cardiac CT and MRI — • Cardiac MRI Protocol
  The cardiac MRI protocol will include cine imaging, aortic flow, and 3D navigator of the aorta. These sequences will be performed to assess aortic root dimensions, including aortic root, sinuses of Valsalva, and sinotubular junction and ascending aorta diameters.
  • CT Aortography Protocol:
  The CT aortography protocol will include non-contrast and contrast-enhanced CT imaging. The non-contrast images will be used for calcium scoring, while the contrast-enhanced images will be used to assess aortic root dimensions

SUMMARY:
Patients who underwent Ross procedure with loose jacket technique will be enrolled in this study and undergo CT and MRI follow-up to compare between both modalities.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent Ross procedure with loose jacket technique at Aswan Heart Centre, regardless of the indication and duration after surgery.
* Patients should have survived until discharge and underwent at least one echocardiography with full data related to one or more anatomic subcomponents of the aortic root before surgery.

Exclusion Criteria:

* Patients who have contraindication for conducting cardiac CT scan. For instance, dye sensitivity, pregnancy, CKD, in addition to patients who have factors that interfere with CT image quality as metallic objects within the chest (e.g. Pacemaker).
* Patients who have contra-indication for conducting a safe MRI scan. For instance, metallic implants that are incompatible with MRI.
* Patients who underwent Ross procedure with technique other than loose jacket.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All paients who underwent Ross procedure with loose jacket technique at Aswan Heart Centre
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MRI measurements in comparison to CT using statistical analysis. | 1 year
  We will use bland altman plots to visualize the degree of agreement between the two raters and identify any systematic bias. The closer the difference to zero, the better.

SECONDARY OUTCOMES:
The largest diameters of each aortic structure | 1 year
  The largest diameters of each aortic structure will be re-calculated as z-scores. In our study, "significant dilatation of the aortic structures" is defined as 95% confidence interval (z-score≥2) in diameter of each aortic structures.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Gamal Ahmed G. Ramadan, Principal Investigator — Assiut University
Locations (1):
- Aswan Heart Centre (Magdi Yacoub Foundation), Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artemiou P, Schusterova I, Tohatyova A, Cocherova J, Krcho P, Sabol F. Follow-up after the Ross procedure, how significant it is, case reports of three patients. J Cardiothorac Surg. 2015 Nov 3;10:144. doi: 10.1186/s13019-015-0369-8. PMID 26530243
- [Background] Ruzmetov M, Welke KF, Geiss DM, Buckley K, Fortuna RS. Failed autograft after the ross procedure in children: management and outcome. Ann Thorac Surg. 2014 Jul;98(1):112-8. doi: 10.1016/j.athoracsur.2014.02.038. Epub 2014 Apr 12. PMID 24725835
- [Background] Juthier F, Vincentelli A, Pincon C, Banfi C, Ennezat PV, Marechaux S, Prat A. Reoperation after the Ross procedure: incidence, management, and survival. Ann Thorac Surg. 2012 Feb;93(2):598-604; discussion 605. doi: 10.1016/j.athoracsur.2011.06.083. Epub 2011 Oct 8. PMID 21983074
- [Background] Notenboom ML, Melina G, Veen KM, De Robertis F, Coppola G, De Siena P, Navarra EM, Gaer J, Ibrahim MEK, El-Hamamsy I, Takkenberg JJM, Yacoub MH. Long-Term Clinical and Echocardiographic Outcomes Following the Ross Procedure: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2024 Jan 1;9(1):6-14. doi: 10.1001/jamacardio.2023.4090. PMID 37938855
- [Background] Notenboom ML, Schuermans A, Etnel JRG, Veen KM, van de Woestijne PC, Rega FR, Helbing WA, Bogers AJJC, Takkenberg JJM. Paediatric aortic valve replacement: a meta-analysis and microsimulation study. Eur Heart J. 2023 Sep 7;44(34):3231-3246. doi: 10.1093/eurheartj/ehad370. PMID 37366156
- [Background] Afifi A, Hosny H, Mahgoub A, Yacoub M. The Ross procedure-the loose jacket technique. Ann Cardiothorac Surg. 2021 Jul;10(4):544-545. doi: 10.21037/acs-2020-rp-20. No abstract available. PMID 34422572
- [Background] Yacoub MH, Tsang V, Sarathchandra P, Jensen H, Hughes S, Latif N. Long-term adaptive versus maladaptive remodelling of the pulmonary autograft after the Ross operation. Eur J Cardiothorac Surg. 2020 May 1;57(5):977-985. doi: 10.1093/ejcts/ezaa019. PMID 32129834
- [Background] Yacoub MH, Notenboom ML, Melina G, Takkenberg JJM. Surgical Heritage: You Had to Be There, Ross: The Comeback Kid. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2024;27:37-41. doi: 10.1053/j.pcsu.2023.10.001. Epub 2023 Nov 7. PMID 38522870
- [Background] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Background] Poskaite P, Pamminger M, Kranewitter C, Kremser C, Reindl M, Reiter G, Piccini D, Dumfarth J, Henninger B, Tiller C, Holzknecht M, Reinstadler SJ, Klug G, Metzler B, Mayr A. Self-navigated 3D whole-heart MRA for non-enhanced surveillance of thoracic aortic dilation: A comparison to CTA. Magn Reson Imaging. 2021 Feb;76:123-130. doi: 10.1016/j.mri.2020.12.003. Epub 2020 Dec 9. PMID 33309920
- [Background] Colan SD, McElhinney DB, Crawford EC, Keane JF, Lock JE. Validation and re-evaluation of a discriminant model predicting anatomic suitability for biventricular repair in neonates with aortic stenosis. J Am Coll Cardiol. 2006 May 2;47(9):1858-65. doi: 10.1016/j.jacc.2006.02.020. Epub 2006 Apr 17. PMID 16682313
- [Background] Gautier M, Detaint D, Fermanian C, Aegerter P, Delorme G, Arnoult F, Milleron O, Raoux F, Stheneur C, Boileau C, Vahanian A, Jondeau G. Nomograms for aortic root diameters in children using two-dimensional echocardiography. Am J Cardiol. 2010 Mar 15;105(6):888-94. doi: 10.1016/j.amjcard.2009.11.040. PMID 20211339
- [Background] Mohammed AFA, Frick M, Kerst G, Hatam N, Elgamal MF, Essa KM, Hovels-Gurich HH, Vazquez-Jimenez JF, Zayat R. Proximal Aortic Dilatation and Pulmonary Valve Replacement in Patients with Repaired Tetralogy of Fallot: Is There a Relationship? A Cardiac Magnetic Resonance Imaging Study. J Clin Med. 2021 Nov 15;10(22):5296. doi: 10.3390/jcm10225296. PMID 34830578